CLINICAL TRIAL: NCT01141686
Title: Non Small Cell Lung Cancer Evaluation According to Pre-determined Drug-targeting Tumor Markers
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Hsingjin Eugene Liu, MD PhD, Taipei Medical University WanFang Hospital
Other Study IDs: IRB98021
Record Dates: First submitted 2010-06-08; First posted 2010-06-10 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluate chemotherapy related tumor markers on non small cell lung cancer by fluorescent in situ hybridization and immunohistochemistry, targets to be studied include EGFR, c-MET, topoisomerase II, p53, topoisomerase I, thymidylate synthase, ERCC1, tau, c-myc, RRM1, class III tubulin. These targets have been chosen because they are targets for chemotherapeutic agents that are currently used in clinical management of these diseases. In total 50 specimen will be studied, approximately one third have mutations/deletions of the EGFR gene.To attempt to establish a correlation between the pre-selected tumor markers and response to chemotherapy, and thus to be able to create a clinically useful classification that would provide clinical guidance for selection of the most effective chemotherapy for a individual patient, and thus be able to logically design more effective clinical trials for the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed lung cancer who received standard platinum-containing doublet chemotherapy followed by EGFR tyrosine kinase inhibitors.

Exclusion Criteria:

* non

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: lung cancer patient in wanfang hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Gjin Eugene Liu, Principal Investigator — Taipei Medical University WanFang Hospital